CLINICAL TRIAL: NCT01361074
Title: In Vivo Versus Augmented Reality Exposure for Small Animal Phobia Treatment: A Randomized Controlled Trial
Brief Title: In Vivo Versus Augmented Reality Exposure for Small Animal Phobia
Acronym: VARESAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UJaumeI01
Record Dates: First submitted 2011-04-26; First posted 2011-05-26 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-09

CONDITIONS: Phobic Disorders
Keywords: Virtual reality; Augmented reality; In vivo exposure; One session treatment; ICT; Efficacy; Specific phobia; Anxiety disorders
MeSH Terms: conditions — Phobic Disorders; Phobia, Specific; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- In Vivo Exposure (Experimental)
  Interventions: Behavioral: In Vivo Exposure for Animal Phobia following Öst´s guidelines
- Augmented Reality Exposure (Experimental)
  Interventions: Behavioral: Augmented Reality Exposure for Animal Phobia following Öst´s guidelines

INTERVENTIONS:
Behavioral: In Vivo Exposure for Animal Phobia following Öst´s guidelines — In vivo exposure is applied using "one-session treatment" guidelines (Öst, Salkovskis and Hellström, 1991). Exposure is conducted in a single extended session lasting up to 3 hours and implemented individually. The treatment includes participant modelling, in vivo exposure, reinforced practice and cognitive challenge. Treatment in a single session is just a starting point; it is recommended that the participants continue to be exposed to the phobic situations after therapy in their daily lives in order to fully surmount their problems. Participants are informed that the treatment required close collaboration between themselves and the therapist. The exposure session is completed in a gradual and planned way.
  Other Names: In vivo exposure in phobic disorders; In vivo exposure for small animal phobia
  Arms: In Vivo Exposure
Behavioral: Augmented Reality Exposure for Animal Phobia following Öst´s guidelines — Augmented Reality (AR) is a variation of Virtual Reality in which the user sees the real world augmented by various virtual elements; it complements reality rather than replacing it completely (Azuma et al., 2001). The most significant aspect of AR is that the virtual elements add relevant and helpful information to the physical information available in the real world. The system includes the options of changing the number, movement and size of small animals. Preliminary data show the utility of the system for the treatment of insect phobia (Botella et al., 2005). AR exposure is applied in the same way than in vivo exposure, that is, in a gradual, planned and controlled way using "one-session treatment" guidelines (Öst, Salkovskis and Hellström, 1991). The therapist can see what the participant sees in AR on a monitor and observe the same stimuli.
  Other Names: Augmented Reality Exposure in phobic disorders; Augmented Reality Exposure for small animal phobia
  Arms: Augmented Reality Exposure

SUMMARY:
The aim of this study is to explore the differential efficacy of in vivo exposure versus augmented reality exposure in the treatment of specific phobia (small animals).

The hypothesis is: There will not be significant statistical differences in the efficacy of in vivo exposure therapy versus augmented reality exposure in the treatment of specific phobia (small animals).

DETAILED DESCRIPTION:
Among anxiety disorders, specific phobias are highly prevalent (around 7.2% and 11.3% in the general population). Cockroach or spider phobia is a type of specific phobia, animal type. The gold standard for the treatment of specific phobia (included small animal phobia) is in vivo exposure. Most phobia sufferers (60-80%) never seek treatment. Besides, not all patients benefit from in vivo exposure, given that an important amount of them do not accept the intervention or drop out (around 25%) when they are informed about the intervention procedure.

Information and Communication Technologies (ICT) like Virtual Reality (VR) and Augmented Reality (AR) are pioneer applications that can improve treatment adherence and acceptance. There exist some studies offering preliminary evidence of the efficacy of AR for the treatment of small animal phobia. However, there are not any controlled study exploring the differential efficacy of ICT-based exposure interventions versus in vivo exposure. In the present study the differential efficacy of AR exposure versus in vivo exposure for the treatment of small animal phobia is explored with a between subject randomized controlled trial. A pre-treatment assessment will be conducted in order to establish the diagnosis and evaluate the main outcome measures. All participants will receive an intensive exposure session following Öst guidelines, (in vivo exposure in one experimental condition and AR exposure in the other experimental condition). After the treatment a post-treatment assessment will be carried out as well as follow-up assessments at 3- and 12-month after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18-65 years of age.
* To meet current DSM-IV-TR criteria for specific phobia (animal type)
* Have as the major presenting complaint anxiety in, and avoidance of, a large range of situations involving spiders or cockroaches.
* A minimum of 1 year duration of the phobia.
* To have scores over 4 in phobic avoidance (on a scale of 0 to 8).
* Express a willingness to participate in the study.

Exclusion Criteria:

* To be able to put a hand inside the container with a spider or cockroach during the behavioral test.
* Have other psychiatric problem in immediate need of treatment.
* Have psychotic or organic symptoms.
* Have heart or lung disease.
* Current alcohol or drug dependence or medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in Behavioral Avoidance Test (BAT, Öst, Salkovskis, and Hellström's, 1991) at pre, post intervention and 3 and 12-month follow-up periods | At pre (baseline), post intervention and 3 and 12-month follow-up periods
  The BAT assesses the severity of the subjective fear, avoidance, and belief in the catastrophic thoughts of the participants on a scale of 0 to 10 before they entered in a room with a feared insect. A container with a live cockroach or spider in it was placed 5 meters from the entrance. Participants were asked to enter the room and approach the insect as closely as possible. They were told that they could terminate the behavioral test at any point. Their performances in the test were scored, taking into account their final proximity to the insect and was converted to a behavioral score.

SECONDARY OUTCOMES:
Change in Spider Phobia Beliefs Questionnaire (SPBQ; adapted from Arntz, Lavy, Van der Berg, & Van Rijsoort, 1993) at pre, post intervention and 3 and 12-month follow-up periods | At pre (baseline), post intervention and 3 and 12-month follow-up periods
  This is a self-report scale with two subscales: items 1-42 assess the strength of fearful beliefs about spiders; items 43-78 measure the strength of fearful beliefs about one's reaction to encountering spiders. Items are rated from 0 to 100. Good internal consistency for both subscales (α=.94) and acceptable test-retest reliability (r=.68 for the spider-related and r=.71 for the self-related one) have been reported. An adaptation of this questionnaire was made by our research team in order to assess fearful beliefs about cockroaches and has been used in other studies (Botella et al., 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Botella, Full Professor, Study Director — University Jaume I, Castellon, Spain.; Cristina Botella, Full Professor, Study Director — University Jaume I, Castellon, Spain
Locations (2):
- Spain (2):
  - University Jaume I, Castellon, Castellon
  - University Jaume I, Castellon, Castellón

REFERENCES:
- [Background] Botella C, Breton-Lopez J, Quero S, Banos R, Garcia-Palacios A. Treating cockroach phobia with augmented reality. Behav Ther. 2010 Sep;41(3):401-13. doi: 10.1016/j.beth.2009.07.002. Epub 2010 Mar 20. PMID 20569788
- [Background] Essau CA, Conradt J, Petermann F. Frequency, comorbidity, and psychosocial impairment of specific phobia in adolescents. J Clin Child Psychol. 2000 Jun;29(2):221-31. doi: 10.1207/S15374424jccp2902_8. PMID 10802831
- [Background] Magee WJ, Eaton WW, Wittchen HU, McGonagle KA, Kessler RC. Agoraphobia, simple phobia, and social phobia in the National Comorbidity Survey. Arch Gen Psychiatry. 1996 Feb;53(2):159-68. doi: 10.1001/archpsyc.1996.01830020077009. PMID 8629891
- [Background] Garcia-Palacios A, Botella C, Hoffman H, Fabregat S. Comparing acceptance and refusal rates of virtual reality exposure vs. in vivo exposure by patients with specific phobias. Cyberpsychol Behav. 2007 Oct;10(5):722-4. doi: 10.1089/cpb.2007.9962. PMID 17927544
- [Background] Garcia-Palacios A, Hoffman HG, See SK, Tsai A, Botella C. Redefining therapeutic success with virtual reality exposure therapy. Cyberpsychol Behav. 2001 Jun;4(3):341-8. doi: 10.1089/109493101300210231. PMID 11710258
- [Background] Marks IM, Mathews AM. Brief standard self-rating for phobic patients. Behav Res Ther. 1979;17(3):263-7. doi: 10.1016/0005-7967(79)90041-x. No abstract available. PMID 526242
- [Background] Botella CM, Juan MC, Banos RM, Alcaniz M, Guillen V, Rey B. Mixing realities? An application of augmented reality for the treatment of cockroach phobia. Cyberpsychol Behav. 2005 Apr;8(2):162-71. doi: 10.1089/cpb.2005.8.162. PMID 15938656
- [Background] Juan MC, Alcaniz M, Monserrat C, Botella C, Banos RM, Guerrero B. Using augmented reality to treat phobias. IEEE Comput Graph Appl. 2005 Nov-Dec;25(6):31-7. doi: 10.1109/mcg.2005.143. No abstract available. PMID 16315475
- [Background] Ost LG. One-session treatment for specific phobias. Behav Res Ther. 1989;27(1):1-7. doi: 10.1016/0005-7967(89)90113-7. PMID 2914000
- [Background] Ost LG. [One-session treatment of specific phobias--a rapid and effective method]. Lakartidningen. 1988 Mar 30;85(13):1139-42. No abstract available. Swedish. PMID 3352391
- See also: Information about our research group — http://www.labpsitec.uji.es/esp/index.php
- See also: International research group that focuses on virtual reality and analgesic effects — http://www.hitl.washington.edu/projects/magnet/